CLINICAL TRIAL: NCT06139913
Title: Effect of Fat Burning Zone of Aerobic Exercise on Fitness Score and Blood Glucose Level in Adolescents Girls With Diabetes Mellitus
Brief Title: Aerobic Exercise on Fitness Score and Blood Glucose Level in Adolescents Girls With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Rana Nabil Hussein Mohamed, Lecturer of pediatric physical therapy in MTIU, MTI University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/2111/MTI.PT2303124
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: prospective study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- aerobic exercise (Experimental): aerobic exercise using treadmill
  Interventions: Other: aerobic exercise

INTERVENTIONS:
Other: aerobic exercise — moderate intensity aerobic exercise using treadmill

SUMMARY:
In adolescent diabetic girls, a correct life style, including diet and physical activity, is part of a correct intervention protocol. Thus, the aim of this study was to evaluate the effects of aerobic training intervention, based on heart rate at glycemic level , on clinical and physiological parameters in adolescent girls with type 1 diabetes forty type1 DM girls will randomly assigned to an intervention (study group ) or control group. The study group will perform a supervised aerobic exercise training based on heart rate whereas control group maintained their usual lifestyle. Anthropometric fitness score measures, blood analysis will assess at baseline and after intervention.

DETAILED DESCRIPTION:
fourty adolescents girls were diagnosed by physician as having type 1 diabetes mellitus and recruited from outpatient internal of El-Hussien hospital in Egypt . girls ages were between 13 and 18yr old; . The following inclusion criteria was applied to all participants in the study : all girls had type 1DM for more than 3 years, Their dose of insulin intake over 0.4 U/Kg/day, Body mass index (BMI) between 25 and 30 kg/m2 . Moderate-intensity aerobic exercise was defined according to the classification standard of the ACSM, which refers to exercise where the HRR of subjects is 64-76%; the moderate-intensity target heart rate area was set in advance and controlled by heart rate monitor during the intervention, and the menarche was began from 3 to 5 years. The patients had no history of severe and frequent hypoglycemia in the last 6 months (< 60 mg/dl, more than twice a week).

All participants attended a clinic for clinical assessments before and after treatment plane.

1. Body Mass Index (BMI)
2. Fitness score
3. Target Heart Rate
4. Fasting blood samples, post prandial and HbA1c: were taken for the following measurements: glucose.
5. Estradiol blood test

ELIGIBILITY:
Inclusion Criteria:

* All girls had type 1DM for more than 3 years,
* Their didn't of insulin intake over 0.4 U/Kg/day, Body mass index (BMI) between 25 and 30 kg/m2

Exclusion Criteria:

* Diabetes as a secondary condition
* Any known cardiac defects and Macrovascular or microvascular chronical complications.
* Insulin therapy and regulate dietary intake Were followed through diabetes physician.

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-09-17 (Actual)

PRIMARY OUTCOMES:
Fitness score: | 3 month
  2- Fitness score: were assessed by multifrequency bioelectrical impedance analysis (MF-BIA; InBody 3.0, Biospace, Seoul, Korea)
Fasting blood samples, post prandial and HbA1c: | 3 month
  Fasting blood samples, post prandial and HbA1c: were taken for the following measurements: glucose.
Estradiol blood test | 3 month
  Estradiol blood test of the participants was done by a laboratory assistant to evaluate the estrogen level of the participants' pre- and post-exercise intervention. The serum concentrations of estradiol (E2) were analyses were performed on day 3 after onset of menstruation

CONTACTS AND LOCATIONS:
Overall Officials: karim sami ibrahim, doctoral, Study Director — lecturer of pediatric physical therapy
Locations (1):
- faculty of pysical therapy, MTI university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No